CLINICAL TRIAL: NCT05680753
Title: A Stratified Approach Integrated With eHealth in Primary Care Physiotherapy for Patients With Neck and/or Shoulder Complaints
Brief Title: Stratified Physiotherapeutic (Blended) Care in Neck and Shoulder Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark van Tilburg (Other)
Responsible Party: Sponsor-Investigator, Mark van Tilburg, Investigator, University of Applied Sciences Utrecht
Organization: University of Applied Sciences Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL69963.041.19; NL8249 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain; Shoulder Pain
Keywords: Stratified care; Physiotherapy; Blended care
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A multicenter, pragmatic, two-arm, parallel-group, cluster randomized controlled trial (cRCT) will be conducted.
Masking Description: Due to the nature of the intervention, blinding of participating physiotherapists is not possible. However, neither physiotherapists nor patients in the usual physiotherapy care arm will be informed about the Stratified Blended Approach arm.
  During the analyses, the researchers will be blinded to group allocation until the entire analysis will be completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratified Blended Approach arm (Experimental): First, physiotherapists will use two stratification tools to decide the most suitable content and intensity as well as mode of care delivery of primary care physiotherapy. The content and intensity of physiotherapy will be matched to the patient's risk of persistent disabling pain as assessed with the Keele STarT MSK tool. The mode of care delivery of physiotherapy will be matched to the patient's suitability for blended care as assessed using the Dutch Blended Physiotherapy Checklist (i.e. yes or no). Second, physiotherapists will receive two practical tools to provide the matched treatment of the mode of care delivery. If considered suitable for blended care, the patient will receive a blended physiotherapy treatment (e-Exercise), in which a smartphone app with personalized information, exercises and physical activity modules is an integral part of physiotherapy treatment. If patients are considered not to be suitable for blended care, a paper-based workbook will be integrated.
  Interventions: Behavioral: Physiotherapy
- Usual physiotherapy arm (Active Comparator): Patients in the usual physiotherapy arm will be offered usual care (face-to-face or video consults) based upon the recommendations of the guidelines of the Royal Dutch Association for Physiotherapy (KNGF). The clinical guideline for neck pain, recommends categorization in treatment profiles based on: the severity of neck pain, the course of symptoms (normal vs. deviant) and the presence of psychosocial factors that may hinder recovery (yes vs. no). The clinical guideline for complaints of the arm, neck and shoulder recommends categorization in treatment profiles based on the region of complaints indicated as most problematic and the relationship between complaints, disabilities, and limitations in participation. No stratification tools to identify patient subgroups and subsequently match them to a treatment are recommended by the guidelines.
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Physiotherapy — Physiotherapy

SUMMARY:
The aim of this cluster RCT is to investigate the clinical effectiveness of a Stratified Blended Approach for patients with neck and/or shoulder complaints on pain and disability over 9 months, compared to usual physiotherapy care.

Our secondary aims are twofold:

* to investigate the effectiveness of the Stratified Blended Approach for patients with neck and/or shoulder complaints on pain intensity, health-related quality of life, illness perceptions, self-management skills, physical activity, exercise adherence, self-perceived effect and satisfaction at 3 and 9 months, compared to usual physiotherapy care;
* to investigate the cost-effectiveness and cost-utility of the Stratified Blended Approach for patients with neck and/or shoulder complaints, compared to usual physiotherapy care.

In the Stratified Blended Approach arm, physiotherapists will match I) the content and intensity of physiotherapy care to the patient's risk of persistent disabling pain, categorized as low, medium or high (using the Keele STarT MSK Tool) and II) the mode of care delivery to the patient's suitability and willingness to receive blended care. The control arm will receive physiotherapy as usual.

This study is financially supported by the Scientific College Physiotherapy (WCF), part of the Royal Dutch Association for Physiotherapy (KNGF). WCF has no role in study design, data collection and analysis, decision to publish, or preparation of the manuscripts. External peer-review took place during the funding process. The results will be publicly disclosed unreservedly.

DETAILED DESCRIPTION:
Intervention:

According to the Stratified Blended approach, patients will be matched to an appropriate treatment based on their risk of persistent disabling pain (assessed with the Keele STarT MSK Tool - either low, medium or high risk) and their suitability for blended care (assessed with the Dutch Blended Physiotherapy Checklist - either suitable or unsuitable for blended care). Based on patients risk profile, the physiotherapy treatment will be targeted to patients' individual needs. If considered suitable for blended care, the patient will receive a digital and face-to-face blend of physiotherapy treatment (e-Exercise) in which an app with personalized information, exercises and physical activity modules is integrated with face-to-face physiotherapy care. If patients are considered unsuitable for blended care, they will receive an information workbook with similar content as the app will be integrated with face-to-face physiotherapy. The app and the information workbook aims to support adherence to physical activity and exercise recommendations. Content of care was based on the Dutch KNGF Clinical Practice Guidelines for Physiotherapy Neck pain, Complaints of Arm, Neck and Shoulder (CANS) and Subacromial complaints.

Control group:

Usual physiotherapy. Content of care was based on the Dutch KNGF Clinical Practice Guidelines for Physiotherapy Neck pain, Complaints of Arm, Neck and Shoulder (CANS) and Subacromial complaints.

ELIGIBILITY:
Inclusion criteria: Patients with neck and/or shoulder complaints will be recruited within participating physiotherapy practices. In order to be eligible to participate in the data collection for the trial, a patient must meet all of the following criteria:

* consulting for physiotherapy for neck and/or shoulder complaints;
* one of the following physiotherapeutic diagnoses: subacromial complaints, biceps tendinosis, shoulder instability or non-specific musculoskeletal complaints of the neck and/or shoulder (not caused by acute trauma (fracture or rupture) or by any systemic disease);
* 18 years or older;
* sufficient mastery of the Dutch language.

Exclusion criteria: A patient who meets any of the following criteria will not be suitable to take part in the data collection for the trial:

* neck and/or shoulder complaints caused by specific pathology (e.g. shoulder pain with loss of active and passive range of motion (frozen shoulder), vertebral fracture, tendon rupture, Parkinson's disease, hernia nucleus pulposus, cervical stenosis), except for subacromial impingement, biceps tendinosis and shoulder instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Neck pain and disability score (NPAD; for patients with neck pain) | 9 months
  The primary outcome is the combined region-specific pain and disability score over 9 months follow-up, assessed by the Neck Pain and Disability Scale (NPAD) for patients with primarily neck complaints and by the Shoulder Pain and Disability Index (SPADI) for patients with primarily shoulder complaints. A higher total score (0-100 for both outcome measures) indicates increased pain and functional limitations.
Shoulder pain and disability index (SPADI; for patients with shoulder pain) | 9 months
  The primary outcome is the combined region-specific pain and disability score over 9 months follow-up, assessed by the Neck Pain and Disability Scale (NPAD) for patients with primarily neck complaints and by the Shoulder Pain and Disability Index (SPADI) for patients with primarily shoulder complaints. A higher total score (0-100 for both outcome measures) indicates increased pain and functional limitations.

SECONDARY OUTCOMES:
Neck and/or shoulder pain intensity | 3 months
  The average neck and/or shoulder pain intensity in the last week will be measured with an 11-point Numeric Rating Scale (NRS) (0 = no pain; 10 = worst pain imaginable)
Neck and/or shoulder pain intensity | 9 months
  The average neck and/or shoulder pain intensity in the last week will be measured with an 11-point Numeric Rating Scale (NRS) (0 = no pain; 10 = worst pain imaginable)
Health-related quality of life | 3 months
  Health-related quality of life will be measured with the 36-Item Short Form Health Survey (SF-36). The questionnaire consists of eight subscales (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain (over the last 4 weeks) and general health). Scores for each subscale will be calculated (0-100). Higher scores indicate a better health-related quality of life.
Health-related quality of life | 9 months
  Health-related quality of life will be measured with the 36-Item Short Form Health Survey (SF-36). The questionnaire consists of eight subscales (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain (over the last 4 weeks) and general health). Scores for each subscale will be calculated (0-100). Higher scores indicate a better health-related quality of life.
Illness perceptions | 3 months
  Illness perceptions will be measured with the Brief Illness Perception Questionnaire (IPQ-K). This questionnaire is an eight-item scale designed to assess cognitive and emotional representations of illness on an ordinal scale (0-10)
Illness perceptions | 9 months
  Illness perceptions will be measured with the Brief Illness Perception Questionnaire (IPQ-K). This questionnaire is an eight-item scale designed to assess cognitive and emotional representations of illness on an ordinal scale (0-10)
Patients' self-management skills | 3 months
  Patients' self-management skills are assessed with the Dutch version of the short form Patient Activation Measure (PAM13-Dutch). The PAM 13-Dutch is a reliable 13-item instrument and assesses patient (or consumer) self-reported knowledge, skills and confidence for self-management of one's health or chronic condition. The answering categories per item are 4-point Likert scales, ranging from totally disagree to totally agree and 'non applicable'. A higher score (range 1-100) indicates a higher level of self-management.
Patients' self-management skills | 9 months
  Patients' self-management skills are assessed with the Dutch version of the short form Patient Activation Measure (PAM13-Dutch). The PAM 13-Dutch is a reliable 13-item instrument and assesses patient (or consumer) self-reported knowledge, skills and confidence for self-management of one's health or chronic condition. The answering categories per item are 4-point Likert scales, ranging from totally disagree to totally agree and 'non applicable'. A higher score (range 1-100) indicates a higher level of self-management.
Physical activity | 3 months
  Physical activity will be objectively measured with an Actigraph accelerometer. The Actigraph accelerometer is a reliable tool for measuring physical activity in adults. Participants will be instructed to wear the accelerometer on their waist for five consecutive days, except when sleeping, showering, bathing or swimming. Average amount of moderate or vigorous physical activity (MVPA) per day will be calculated.
Physical activity | 9 months
  Physical activity will be objectively measured with an Actigraph accelerometer. The Actigraph accelerometer is a reliable tool for measuring physical activity in adults. Participants will be instructed to wear the accelerometer on their waist for five consecutive days, except when sleeping, showering, bathing or swimming. Average amount of moderate or vigorous physical activity (MVPA) per day will be calculated.
Exercise adherence | 3 months
  Exercise adherence will be measured with the Exercise Adherence Rating Scale (EARS). The EARS is a 6 item self-reported questionnaire with items scored on a 5-point Likert scale (0 = completely agree; 4 = completely disagree). A higher score (0-24) indicates better adherence to prescribed home-exercises.
Exercise adherence | 9 months
  Exercise adherence will be measured with the Exercise Adherence Rating Scale (EARS). The EARS is a 6 item self-reported questionnaire with items scored on a 5-point Likert scale (0 = completely agree; 4 = completely disagree). A higher score (0-24) indicates better adherence to prescribed home-exercises.
Global perceived effect | 3 months
  Global perceived effect will be measured with the 7-point Likert global perceived effect score (GPE). Categories 1 (very much improved) to 3 (a little improved) are classified as 'improved'. Categories 4 (no change) to 7 (very much worse) are classified as 'not improved'.
Global perceived effect | 9 months
  Global perceived effect will be measured with the 7-point Likert global perceived effect score (GPE). Categories 1 (very much improved) to 3 (a little improved) are classified as 'improved'. Categories 4 (no change) to 7 (very much worse) are classified as 'not improved'.
Satisfaction with treatment | 3 months
  Satisfaction with treatment outcome will be measured with an 8-point Likert scale question: 'All things considered, how satisfied are you with the results of the treatment for your neck and/or shoulder complaints? (1 = extremely satisfied, 7 = extremely dissatisfied, 8 = not sure/no opinion)
Neck pain and disability score (NPAD; for patients with neck pain) | 3 months
  This outcome will be combined to a region-specific pain and disability score over 3 months follow-up, assessed by the Neck Pain and Disability Scale (NPAD) for patients with primarily neck complaints and by the Shoulder Pain and Disability Index (SPADI) for patients with primarily shoulder complaints. A higher total score (0-100 for both outcome measures) indicates increased pain and functional limitations.
Shoulder pain and disability index (SPADI; for patients with shoulder pain) | 3 months
  This outcome will be combined to a region-specific pain and disability score over 3 months follow-up, assessed by the Neck Pain and Disability Scale (NPAD) for patients with primarily neck complaints and by the Shoulder Pain and Disability Index (SPADI) for patients with primarily shoulder complaints. A higher total score (0-100 for both outcome measures) indicates increased pain and functional limitations.
Cost-effectiveness (assessed with a cost questionnaire) | 9 months
  A cost-utility analysis (CUA) will be performed for QALYs and a cost-effectiveness analysis (CEA) for the combined region-specific pain and disability score, both of which will be performed from the societal and the healthcare perspective. From the societal perspective all costs will be taken into account, irrespective of who pays or benefits, whereas solely those borne by the healthcare sector will be included if the healthcare perspective is applied.
Cost-utility (assessed with a cost questionnaire) | 9 months
  A cost-utility analysis (CUA) will be performed for QALYs and a cost-effectiveness analysis (CEA) for the combined region-specific pain and disability score, both of which will be performed from the societal and the healthcare perspective. From the societal perspective all costs will be taken into account, irrespective of who pays or benefits, whereas solely those borne by the healthcare sector will be included if the healthcare perspective is applied.

OTHER OUTCOMES:
The content of physiotherapy care | Through treatment completion, an average of 3 months
  The content and intensity of physiotherapy care will be measured by a case report form, filled out by the physiotherapist at the end of the treatment period or after 3 months. Information of the risk of persistent disabling pain, the suitability for blended care, the physiotherapists diagnosis of the presenting problem, the number of physiotherapy sessions, deviations from the study protocol, and content of the physiotherapy sessions will be collected.
The intensity of physiotherapy care | Through treatment completion, an average of 3 months
  The content and intensity of physiotherapy care will be measured by a case report form, filled out by the physiotherapist at the end of the treatment period or after 3 months. Information of the risk of persistent disabling pain, the suitability for blended care, the physiotherapists diagnosis of the presenting problem, the number of physiotherapy sessions, deviations from the study protocol, and content of the physiotherapy sessions will be collected.
Adherence to the smartphone app with e-Exercise modules in the Stratified Blended Approach arm | Through treatment completion, an average of 3 months
  Adherence to the smartphone app with e-Exercise modules in the Stratified Blended Approach arm will be assessed by quantitative data on the usage. These data will automatically be stored on the backend of the app.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Veenhof, Prof. dr., Principal Investigator — HU University of applied sciences Utrecht
Locations (1):
- HU University of applied sciences Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: SAP
Time Frame: Data will first be used by the research team for analyses. Then we will determine when data will be made available. Within the limitations of protecting personal data, we strive to make the datasets and syntaxes as openly available as possible to ensure the transparency and reproducibility of our research.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT05680753/SAP_000.pdf